CLINICAL TRIAL: NCT04996394
Title: Effects of Neuromuscular Blocking Agents on End Expiratory Lung Volume During Moderate-severe ARDS
Brief Title: "Effects of Neuromuscular Blocking Agents on End Expiratory Lung Volume During Moderate-severe ARDS"
Acronym: EIT_CURARO
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: EIT_CURARO
Record Dates: First submitted 2021-04-03; First posted 2021-08-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: ARDS; Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMBAs

SUMMARY:
This is a monocentric, prospective, observational study that will be conducted in the general ICU of San Gerardo Hospital (Monza, Italy). Study protocol will be started when NMBAs infusion will be stopped for clinical reason until regain of spontaneous breathing activity.

Patients will be enrolled at the moment of NMBAs infusion interruption ("baseline" phase). Clinical data will be collected: hemodynamics, ventilation parameters and respiratory mechanics, arterial blood gas analysis, drugs used for sedation and their dosages. An EIT belt will be positioned around the patient's chest when clinical signs of spontaneous breathing activity will be detectable (unstable flow curve on the ventilator, deflection in airway pressure during an expiratory pause). In this phase ("NMBA interruption") same clinical data will be collected as at baseline. Patients will be ventilated in the same ventilation mode as before (Volume Controlled mechanical ventilation), but the inspiratory trigger on the ventilator will be turned on to reduce patient-ventilator asynchronies. When an EIT trace lasting at least 10 minutes will be recorded, an NMBA bolus (as prescribed by the treating physician) will be administered and a continuous infusion will be restarted. Clinical data will be collected again in this phase ("NMBA restart").

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate-severe ARDS (according to Berlin definition)
* Patients treated with NMBAs
* age>18 years old

Exclusion Criteria:

* pregnancy,
* presence of air leaks (ex. presence of broncho-pleural fistula or pneumothorax)
* presence of contraindications to EIT belt positioning ( ex. presence of pace-makers, presence of unstable spinal fractures).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-severe ARDS (according to Berlin definition) needing NMBAs administration will be included
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
End Expiratory Lung Volume | Entire study duration (approx. 1 year)
  Patients will be enrolled at the moment of NMBAs infusion interruption ("baseline" phase). An EIT belt will be positioned around the patient's chest when clinical signs of spontaneous breathing activity will be detectable (unstable flow curve on the ventilator, deflection in airway pressure during an expiratory pause). In this phase ("NMBA interruption") same clinical data will be collected as at baseline. When an EIT trace lasting at least 10 minutes will be recorded, an NMBA bolus (as prescribed by the treating physician) will be administered and a continuous infusion will be restarted. Clinical data will be collected again in this phase ("NMBA restart").

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza, Monza, Lombardy, Italy

REFERENCES:
- [Background] Murray MJ, DeBlock H, Erstad B, Gray A, Jacobi J, Jordan C, McGee W, McManus C, Meade M, Nix S, Patterson A, Sands MK, Pino R, Tescher A, Arbour R, Rochwerg B, Murray CF, Mehta S. Clinical Practice Guidelines for Sustained Neuromuscular Blockade in the Adult Critically Ill Patient. Crit Care Med. 2016 Nov;44(11):2079-2103. doi: 10.1097/CCM.0000000000002027. PMID 27755068
- [Background] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- [Background] Gainnier M, Roch A, Forel JM, Thirion X, Arnal JM, Donati S, Papazian L. Effect of neuromuscular blocking agents on gas exchange in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2004 Jan;32(1):113-9. doi: 10.1097/01.CCM.0000104114.72614.BC. PMID 14707568
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Fanelli V, Morita Y, Cappello P, Ghazarian M, Sugumar B, Delsedime L, Batt J, Ranieri VM, Zhang H, Slutsky AS. Neuromuscular Blocking Agent Cisatracurium Attenuates Lung Injury by Inhibition of Nicotinic Acetylcholine Receptor-alpha1. Anesthesiology. 2016 Jan;124(1):132-40. doi: 10.1097/ALN.0000000000000907. PMID 26540149
- [Background] Forel JM, Roch A, Marin V, Michelet P, Demory D, Blache JL, Perrin G, Gainnier M, Bongrand P, Papazian L. Neuromuscular blocking agents decrease inflammatory response in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2006 Nov;34(11):2749-57. doi: 10.1097/01.CCM.0000239435.87433.0D. PMID 16932229
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Background] Guervilly C, Bisbal M, Forel JM, Mechati M, Lehingue S, Bourenne J, Perrin G, Rambaud R, Adda M, Hraiech S, Marchi E, Roch A, Gainnier M, Papazian L. Effects of neuromuscular blockers on transpulmonary pressures in moderate to severe acute respiratory distress syndrome. Intensive Care Med. 2017 Mar;43(3):408-418. doi: 10.1007/s00134-016-4653-4. Epub 2016 Dec 24. PMID 28013329